CLINICAL TRIAL: NCT04039451
Title: Prevalence of Psoriasis and Vitiligo in Assiut Governorate, Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aml Hassan Ali, principal investigator, Assiut University
Other Study IDs: POPAVIassiutGE
Record Dates: First submitted 2019-07-16; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Psoriasis; Vitiligo
MeSH Terms: conditions — Psoriasis; Vitiligo

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- people who live in rural areas in Assuit governorate: The study will performed on people who live in rural areas in Assuit governorate (all households) regardless of sex or age.

SUMMARY:
Psoriasis is a chronic, immune-mediated inflammatory skin disease, which ranges in severity from a few scattered red, scaly plaques to involvement of almost the entire body surface. It may progressively worsen with age, or wax and wane in its severity; the degree of severity depends on inheritance and environmental factors.

It is a complex disease, multiple exogenous and endogenous stimuli incite already stimulated innate immune responses in genetically predetermined individuals. The disease process is a result of a network of cell types including T cells, dendritic cells and keratinocytes that, with the production of cytokines, generate a chronic inflammatory state.

Vitiligo is a chronic disorder of pigmentation characterized by the development of white macules on the skin due to loss of epidermal melanocytes.

Its pathogenesis is still unclear, many mechanisms and theories have been suggested including autoimmunity, auto cytotoxicity, biochemical and neuronal mechanisms.

DETAILED DESCRIPTION:
There are multiple patterns of psoriasis including plaque, guttate, pustular, inverse and erythrodermic, approximately 80% of patients present with plaque psoriasis which is clinically characterized by well demarcated erythematous plaques with overlying scales. These plaques can be intensely pruritic and bleed when manipulated, referred to as the Auspitz sign. Lesions are usually distributed symmetrically and frequently occur on the elbows, knees, lower back and scalp.

Prevalence of psoriasis is around 2-3% of the general population. A high prevalence of psoriasis at the rate of 11.8% has been reported from Kazach'ye, located in the Arctic region of the former Soviet Union.

In Egypt, the prevalence reported is around 3%. A study was done in hospitals of Damietta governorate reveals that prevalence of psoriasis is about 5%. Up to the investigator's knowledge the prevalence of psoriasis at Assuit governorate is not known till now.

Vitiligo can be classified into segmental or non-segmental. Non-segmental or generalized vitiligo is the most common clinical presentation and often involves the face and acral regions.

Prevalence of vitiligo is 0.5%-2% of general population world-wide, without predilection for sex or race. A previous study on skin diseases I Assiut governorates reveals that prevalence of vitiligo was about 1.22%.

ELIGIBILITY:
Inclusion Criteria:

* The study will performed on people who live in rural areas in Assuit governorate (all households) regardless of sex or age.

Exclusion Criteria:

* no exclusion criteria

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will performed on people who live in rural areas in Assuit governorate (all households) regardless of sex or age.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-02-29 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of psoriasis and vitiligo in Assuit governorate | 6 months
  Complete history will be obtained from patients: including name, age, sex, occupation, marital status, special habits and risk factors of psoriasis and vitiligo, including history of psoriasis and vitiligo (onset, course, duration, precipitating and previous treatments).

SECONDARY OUTCOMES:
Find the possible precipitating factors affecting. | 2 months
  obtained from history of what exaggerate or decrease the disease.
Types of psoriasis and vitiligo in Assiut governorate | 2 months
  Dermatological examination will be done to find the distribution and extent of the diseases to determine the types.
Severity of psoriasis in Assiut patients | 2 months
  Scoring system will be fulfilled:- Psoriasis area and severity index.
Impact of psoriasis and on Assiut patients | 2 months
  Questionnaire will be fulfilled:- Quality of life of psoriasis patients.
Severity of vitiligo in Assiut patients | 2 months
  Scoring system will be fulfilled:- Vitiligo area severity index score.
Impact of vitiligo and on Assiut patients | 2 months
  Questionnaire will be fulfilled:- Quality of life of vitiligo patients.
Extent of vitiligo | 2 months
  Scoring system will be fulfilled:- vitiligo extent score
Finding associated comorbidities | 2 months
  general examination including joint examination to find associated diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parisi R, Symmons DP, Griffiths CE, Ashcroft DM; Identification and Management of Psoriasis and Associated ComorbidiTy (IMPACT) project team. Global epidemiology of psoriasis: a systematic review of incidence and prevalence. J Invest Dermatol. 2013 Feb;133(2):377-85. doi: 10.1038/jid.2012.339. Epub 2012 Sep 27. PMID 23014338
- [Background] Lebwohl M. Psoriasis. Lancet. 2003 Apr 5;361(9364):1197-204. doi: 10.1016/S0140-6736(03)12954-6. PMID 12686053
- [Background] Nestle FO, Kaplan DH, Barker J. Psoriasis. N Engl J Med. 2009 Jul 30;361(5):496-509. doi: 10.1056/NEJMra0804595. No abstract available. PMID 19641206
- [Background] Finlay AY, Khan GK, Luscombe DK, Salek MS. Validation of Sickness Impact Profile and Psoriasis Disability Index in Psoriasis. Br J Dermatol. 1990 Dec;123(6):751-6. doi: 10.1111/j.1365-2133.1990.tb04192.x. PMID 2265090
- [Background] Raychaudhuri SP, Farber EM. The prevalence of psoriasis in the world. J Eur Acad Dermatol Venereol. 2001 Jan;15(1):16-7. doi: 10.1046/j.1468-3083.2001.00192.x. No abstract available. PMID 11451313
- [Background] Ezzedine K, Eleftheriadou V, Whitton M, van Geel N. Vitiligo. Lancet. 2015 Jul 4;386(9988):74-84. doi: 10.1016/S0140-6736(14)60763-7. Epub 2015 Jan 15. PMID 25596811
- [Background] Salah Eldin MM, Sami NA, Aly DG, Hanafy NS. Comparison Between (311-312 nm) Narrow Band Ultraviolet-B Phototherapy and (308 nm) Monochromatic Excimer Light Phototherapy in Treatment of Vitiligo: A Histopathological Study. J Lasers Med Sci. 2017 Summer;8(3):123-127. doi: 10.15171/jlms.2017.22. Epub 2017 Jun 27. PMID 29123631
- [Background] Alikhan A, Felsten LM, Daly M, Petronic-Rosic V. Vitiligo: a comprehensive overview Part I. Introduction, epidemiology, quality of life, diagnosis, differential diagnosis, associations, histopathology, etiology, and work-up. J Am Acad Dermatol. 2011 Sep;65(3):473-491. doi: 10.1016/j.jaad.2010.11.061. PMID 21839315
- [Background] Abdel-Hafez K, Abdel-Aty MA, Hofny ER. Prevalence of skin diseases in rural areas of Assiut Governorate, Upper Egypt. Int J Dermatol. 2003 Nov;42(11):887-92. doi: 10.1046/j.1365-4362.2003.01936.x. PMID 14636205
- [Background] CAPMAS (2018): The Central Agency for Public Mobilization and Statistics (CAPMAS). The Annual Book of National Statistics. Cairo, Egypt: 2018: 8.
- [Background] Fredriksson T, Pettersson U. Severe psoriasis--oral therapy with a new retinoid. Dermatologica. 1978;157(4):238-44. doi: 10.1159/000250839. PMID 357213
- [Background] Robinson A, Kardos M, Kimball AB. Physician Global Assessment (PGA) and Psoriasis Area and Severity Index (PASI): why do both? A systematic analysis of randomized controlled trials of biologic agents for moderate to severe plaque psoriasis. J Am Acad Dermatol. 2012 Mar;66(3):369-75. doi: 10.1016/j.jaad.2011.01.022. Epub 2011 Oct 29. PMID 22041254
- [Background] van Geel N, Lommerts J, Bekkenk M, Wolkerstorfer A, Prinsen CAC, Eleftheriadou V, Taieb A, Picardo M, Ezzedine K, Speeckaert R. Development and Validation of the Vitiligo Extent Score (VES): an International Collaborative Initiative. J Invest Dermatol. 2016 May;136(5):978-984. doi: 10.1016/j.jid.2015.12.040. Epub 2016 Jan 28. PMID 26827762
- [Background] McKenna SP, Cook SA, Whalley D, Doward LC, Richards HL, Griffiths CE, Van Assche D. Development of the PSORIQoL, a psoriasis-specific measure of quality of life designed for use in clinical practice and trials. Br J Dermatol. 2003 Aug;149(2):323-31. doi: 10.1046/j.1365-2133.2003.05492.x. PMID 12932239
- [Background] Marissa D. Newman and Jeffrey M. Weinberg (2008): The pathophysiology of psoriasis: Treatment of psoriasis; 12,19,11-23.
- [Background] Farber EM and Nail L. (1998): Natural history and genetics. Psoriasis, 3rd edn. Marcel Dekker, New York, 1998: 107-157.